CLINICAL TRIAL: NCT03654378
Title: Defining Factors Responsible for Temporal Changes in CYP3A4-Mediated Drug Metabolism During Pregnancy
Brief Title: Molecular Basis of Altered Drug Metabolism During Pregnancy
Status: Withdrawn | Type: Observational
Why Stopped: Limited participants for enrollment
Sponsor: Northwestern University (Other)
Collaborators: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Katherine Wisner, Professor, Northwestern University
Other Study IDs: NICHD-1 R01 HD089455-01A1
Record Dates: First submitted 2018-08-22; First posted 2018-08-31 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Pregnancy
Keywords: Quetiapine; Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

SUMMARY:
The objectives of this application are to provide mechanistic understanding of altered drug metabolism by hepatic cytochrome CYP3A4 and to translate the findings to human pregnancy. A drug metabolized by CYP3A4, Quetiapine, will be the drug of choice mechanism to understand the enzyme's induction. Pregnant women currently on Quetiapine will be recruited. If the women enroll, the women will participate in four pharmacokinetic (PK) studies (one per trimester, and one postpartum).

DETAILED DESCRIPTION:
The purpose of this research is to understand changes in a woman's body during pregnancy, specifically how the body processes medication during pregnancy.

The investigators know that over 90% of women take at least one drug during pregnancy. Because of the changes in a pregnant women's body, processes such as the rate of drug metabolism can change over the course of the three trimesters.

Drug metabolism is sometimes controlled by certain genes in the body. This study will be examining the up-regulation, or "speeding up" of a certain gene called CYP3A4, a gene that helps the body process Quetiapine.

The primary goal of this research is to understand how drug metabolism changes across pregnancy. The secondary goal for this research is to define how enzymes in the liver act to up-regulate CYP3A4 during pregnancy. This research will help to build a knowledge base for the prediction of drug metabolism changes and the design of optimal individualized dosage regimens for pregnant women.

The results of this study are expected to have a positive impact, as they will lay a foundation for the design of individualized drug therapy during pregnancy. This foundation will minimize the risk of over- and under-dosing pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45 years
* Pregnant, prior to 16 weeks gestation
* No chronic diseases or chronically administered medication
* Singleton or multiple gestation
* Subject may take aspirin, folate/multivitamins and other approved concomitant medications
* Taking Quetiapine for any clinical indication during pregnancy and postpartum
* Has made decision for Quetiapine treatment with prescriber prior to study entry

Exclusion Criteria:

* Chronic use of prescription or over the counter durgs during pregnancy with the exceptions listed under inclusions
* Substance dependence in the last 6 months
* Suicidal ideation with intent or suicide attempt in the last 6 months

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Community sample of women taking Quetiapine in areas surrounding Chicago, IL.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in concentration-to-dose ratio of Quetiapine in plasma | Between 12-15 weeks, 22-25 weeks, 32-35 weeks and 12-15 months postpartum.

SECONDARY OUTCOMES:
Change in thyroid hormone levels in plasma | Between 12-15 weeks, 22-25 weeks, 32-35 weeks and 12-15 months postpartum.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine L Wisner, M.D., M.S., Principal Investigator — Northwestern University; Hyunyoung Jeong, PharmD, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- Northwestern University Asher Center for the Study and Treatment of Depressive Disorders, Chicago, Illinois, United States